CLINICAL TRIAL: NCT07392060
Title: A Randomized, Open-Label, Controlled, Multicenter Phase III Clinical Study of WX390 Combined With Toripalimab Versus Investigator's Choice of Therapy in Patients With Recurrent or Metastatic Cervical Cancer Who Have Failed Prior Platinum-Based Treatment
Brief Title: A Phase III Clinical Study of WX390 Combined With Toripalimab Versus Investigator's Choice of Therapy in Patients With Recurrent or Metastatic Cervical Cancer Who Have Failed Prior Platinum-Based Treatment
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiatan Pharmatech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JYP0390M301
Record Dates: First submitted 2026-01-20; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer Metastatic
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WX390 1.1mg + Toripalimab 240mg (Experimental): Participants will receive WX390 continuous oral dosing (1.1 mg once a day) and Toripalimab fixed dose (240mg, intravenous, Day 1, every 3 weeks).
  Interventions: Drug: WX390 1.1mg + Toripalimab 240mg
- Investigator's Choice of Chemotherapy (Active Comparator)
  Interventions: Drug: Investigator's Choice of Chemotherapy

INTERVENTIONS:
Drug: WX390 1.1mg + Toripalimab 240mg — Participants will receive WX390 continuous oral dosing (1.1 mg once a day) and Toripalimab fixed dose (240mg, intravenous, Day 1, every 3 weeks).
  Arms: WX390 1.1mg + Toripalimab 240mg
Drug: Investigator's Choice of Chemotherapy — Randomization for these two strata will be closed upon reaching the total enrollment of 310 subjects who are immunotherapy-naïve or have tumors with PIK3CA wild-type status confirmed by the central laboratory.
  Arms: Investigator's Choice of Chemotherapy

SUMMARY:
This is a Randomized, Open-Label, Controlled, Multicenter Phase III Clinical Study to evaluate the efficacy of WX390 in combination with toripalimab versus investigator's choice of therapy in patients with recurrent or metastatic cervical cancer who have failed at least one prior platinum-based systemic therapy, as assessed by overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily participates in this clinical study, has provided signed informed consent prior to the initiation of any screening procedures, and is able to understand and comply with the study requirements.
2. Aged 18 to 75 years (inclusive, calculated on the day of signing the informed consent form).
3. Histologically or cytologically confirmed cervical cancer, including squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma.
4. Not eligible for curative treatment with surgery, radiotherapy, or chemoradiotherapy.

   Willing to undergo a biopsy during the screening period to provide fresh tumor tissue for PD-L1 and PIK3CA mutation testing; if a biopsy is not feasible, archived tumor tissue samples (formalin-fixed, paraffin-embedded (FFPE) blocks or unstained FFPE slides) may be provided for PD-L1 testing. All testing will be performed at a central laboratory. If the provided tumor tissue sample is deemed unsuitable by the central laboratory for evaluating PD-L1 expression and/or PIK3CA mutation status, the subject cannot be enrolled.
5. Must have at least one measurable lesion as per RECIST v1.1 criteria. Previously irradiated lesions with confirmed progression on imaging may be considered as target lesions.
6. ECOG performance status of 0 or 1.
7. Able to swallow tablets normally.
8. Life expectancy of ≥3 months.

Exclusion Criteria:

1. Previous treatment with any PI3K, AKT, or mTOR inhibitor, or prior treatment with toripalimab.
2. Patients with type 1 or type 2 diabetes mellitus.
3. History of interstitial lung disease, drug-induced pneumonitis, pulmonary fibrosis, pneumoconiosis, or radiation pneumonitis (patients with only radiographic evidence of radiation pneumonitis and not requiring corticosteroid therapy may be enrolled). Patients with active pneumonia during screening, severely impaired lung function, or other conditions that may interfere with the detection and management of suspected drug-related pulmonary toxicity.
4. Radiographic evidence of tumor invasion into the bladder or rectum, deemed by the investigator to pose a risk of perforation; or a known history of female reproductive tract fistula (e.g., vesicovaginal fistula, urethrovaginal fistula, cervicovesical fistula, etc.). Patients may be enrolled if the perforation or fistula has been treated with diversion surgery, resection, or repair, and the condition is considered resolved or controlled by the investigator.
5. Currently active bleeding, intra-abdominal abscess, or intestinal obstruction requiring clinical intervention.
6. CT/MRI or other imaging shows tumor invasion or encasement of major blood vessels, indicating a high risk of bleeding.
7. Current clinically significant hydronephrosis. Patients may be enrolled if hydronephrosis is relieved by nephrostomy or ureteral stent placement.
8. Patients with refractory nausea and vomiting, dysphagia, gastrointestinal disorders affecting drug absorption (e.g., Crohn's disease, ulcerative colitis, or short bowel syndrome), or other malabsorption conditions.
9. History of severe allergy, hypersensitivity, or other anaphylactic reactions to the investigational product or any of its excipients.
10. Administration of a live vaccine within 4 weeks prior to randomization or planned administration during the study.
11. Patients with active autoimmune disease, history of bone marrow or solid organ transplantation, suicidal tendency, alcohol or drug dependence, clear history of neurological or psychiatric disorders, or other conditions that, in the investigator's assessment, may contraindicate the use of the investigational product, compromise the interpretation of study results, or result in forced discontinuation from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival in cervical cancer patients who have failed at least one prior line of platinum-based therapy | through study completion, an average of 3 years

SECONDARY OUTCOMES:
Efficacy including ORR was assessed by both the investigator and a Blinded Independent Central Review committee according to RECIST v1.1 criteria. | through study completion, an average of 1 year
Adverse Events (AEs), including type, incidence, grading (assessed according to the NCI-CTCAE v5.0 criteria), severity, and relationship to the investigational drug, among others. | through study completion, an average of 3 years
Efficacy including DCR was assessed by both the investigator and a Blinded Independent Central Review committee according to RECIST v1.1 criteria. | through study completion, an average of 1 year
Efficacy including DoR was assessed by both the investigator and a Blinded Independent Central Review committee according to RECIST v1.1 criteria. | through study completion, an average of 1 year